CLINICAL TRIAL: NCT00000244
Title: Effects of Dynorphin 1-13 on Heroin Addiction
Brief Title: Effects of Dynorphin 1-13 on Heroin Addiction - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-08067-1; R01DA008067 (NIH); R01-08067-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Opioid-Related Disorders; Substance Withdrawal Syndrome
Keywords: addiction; opiate; heroin; dynorphin
MeSH Terms: conditions — Opioid-Related Disorders; Substance Withdrawal Syndrome; Behavior, Addictive; Spinocerebellar ataxia 23 | interventions — dynorphin (1-13)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Dynorphin 1 - 13

SUMMARY:
The purpose of this study is to evaluate the effects of IV dynorphin in humans during acute heroin abstinence, in order to determine that dynorphin suppresses acute opiate withdrawal, reduces opiate craving, and is safe at doses required to produce the above effects.

DETAILED DESCRIPTION:
Randomized double blinded study of the effects of a single IV dose of dynorphin A 1-13 on heroin withdrawal in human opiate addicts

ELIGIBILITY:
Inclusion Criteria:

opiate addict between the ages of 18-55

Exclusion Criteria:

Regular abuse of other drugs, unstable medical conditions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1994-08; Primary Completion 1997-03 (Actual); Study Completion 1997-03 (Actual)

PRIMARY OUTCOMES:
Craving scale

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pentel, M.D., Principal Investigator — University of Minnesota
Locations (1):
- U of Minnesota School of Medicine, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Specker S, Wananukul W, Hatsukami D, Nolin K, Hooke L, Kreek MJ, Pentel PR. Effects of dynorphin A(1-13) on opiate withdrawal in humans. Psychopharmacology (Berl). 1998 Jun;137(4):326-32. doi: 10.1007/s002130050626. PMID 9676891